CLINICAL TRIAL: NCT03117309
Title: Phase II Study of Front Line Therapy With Nivolumab and Salvage Nivolumab + Ipilimumab in Patients With Advanced Renal Cell Carcinoma. HCRN: GU16-260
Brief Title: Study of Front Line Therapy With Nivolumab and Salvage Nivolumab + Ipilimumab in Patients With Advanced Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael B. Atkins, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor-Investigator, Michael B. Atkins, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU16-260
Record Dates: First submitted 2017-04-10; First posted 2017-04-17 (Actual); Results first posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Advanced Renal Cell Carcinoma
Keywords: Nivolumab; Ipilimumab; OPDIVO; IgG1 kappa immunoglobulin
MeSH Terms: interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PART A: Nivolumab (Experimental): Nivolumab 240mg; Nivolumab 360mg
  Interventions: Drug: Nivolumab 240 mg; Drug: Nivolumab 360mg
- PART B: Nivolumab + Ipilimumab (Experimental): Nivolumab 3mg/kg and Ipilimumab 1mg/kg; Nivolumab 360mg
  Interventions: Drug: Ipilimumab 1mg/kg; Drug: Nivolumab 3mg/kg; Drug: Nivolumab 360mg

INTERVENTIONS:
Drug: Nivolumab 240 mg — PART A Nivolumab 240 mg IV every 2 weeks x 6 then initial disease assessment
  Other Names: OPDIVO
  Arms: PART A: Nivolumab
Drug: Ipilimumab 1mg/kg — Ipilimumab 1 mg/kg every 3 weeks x 4
  Other Names: Yervoy
  Arms: PART B: Nivolumab + Ipilimumab
Drug: Nivolumab 3mg/kg — In combination with Ipilimumab
  Other Names: OPDIVO
  Arms: PART B: Nivolumab + Ipilimumab
Drug: Nivolumab 360mg — Continue Nivolumab 360 mg IV every 3 weeks
  Other Names: OPDIVO

SUMMARY:
Phase II trial of nivolumab in 120 treatment naïve patients with ccRCC.

DETAILED DESCRIPTION:
Eligible patients with biopsiable (biopsied) disease will receive nivolumab 240 mg IV every 2 weeks x 6 doses then 360 mg every 3 weeks for up to 84 weeks. Tumor response will be assessed at weeks 12, 18 and 24 and then every 12 weeks. For patients who experience RECIST 1.1 defined PD, but remain clinically stable (and asymptomatic), a confirmatory scan after 6 weeks (± 1 week) of additional therapy is suggested. Patients with persistent PD at confirmatory scan will be evaluated for enrollment on Part B of this study. Symptomatic patients may be evaluated for Part B immediately. Patients without confirmed PD can continue on nivolumab therapy.

Patients who experience symptomatic or confirmed PD (or have best response of SD at 12 months) on nivolumab monotherapy will be eligible for consideration for Part B. Part B involves the addition of ipilimumab for up to 4 doses while maintaining nivolumab therapy. Dose of ipilimumab will be 1 mg/kg every 3 weeks together with nivolumab changed to 3 mg/kg every 3 weeks for up to 4 doses. Nivolumab will revert to 360 mg every 3 weeks after the completion of treatment with ipilimumab (beginning week 13-19 of Part B) for up to 48 weeks. Patients will be followed with serial imaging assessments weeks 12, 18 and 24 and then every 12 weeks after the initiation of ipilimumab. The tumor measurements at the time of ipilimumab institution will be the new baseline. If unequivocal symptomatic or confirmed new PD (as defined above) develops, treatment will be discontinued.

Patients for Part B must still meet the eligibility criteria for initial study enrollment. Patients with Grade 3 toxicity on nivolumab monotherapy, serious symptomatic disease that in the opinion of the site investigator requires immediate use of an alternative treatment approach or continued PR/CR will be excluded from enrolling in Part B. It is estimated that roughly half of the patients accrued to the first-line treatment will go on to enroll in Part B.

An additional biopsy will be performed of a metastatic lesion at time of confirmed PD in all patients enrolling in Part B. Confirmation of tumor in the biopsy specimen must occur prior to initiation of treatment on Part B. FFPE and frozen tissue will be stored from this sample and used for correlative studies described below.

An additional cohort of 40 non-ccRCC patients will be enrolled and analyzed separately for evidence of anti-tumor activity (CR, PR and SD and PFS at 1 year of nivolumab). These patients will also be eligible for participation in Part B. We anticipate that the accrual of these 40 patients will be able to be completed within the 1.5 years needed for accrual of the ccRCC patients.

Part A: Nivolumab Administration. Nivolumab will be given every 2 weeks x 6 at a dose of 240 mg Intravenously (IV) and then every 3 weeks at a dose of 360 mg IV until toxicity, complete response, disease progression, SD at 12 months or a maximum of 96 total weeks (12 weeks induction, 84 weeks maintenance) Patients with disease progression (at any time) or SD at 12 months will be eligible to be considered for participation in Part B of the study.

Part B: Nivolumab + Ipilimumab. Patients with Grade 3 toxicity on nivolumab monotherapy, (excluding endocrine toxicity), serious symptomatic disease that in the opinion of the site investigator requires immediate use of an alternative treatment approach or continued PR/CR will be excluded from enrolling in Part B. It is estimated that roughly half of the patients accrued to the first line treatment will go on to enroll in Part B.

Ipilimumab will be given 1 mg/kg every 3 weeks together with nivolumab 240 mg every 3 weeks for up to 4 doses. Nivolumab will revert to 3 mg/kg every 3 weeks after the completion of combination treatment with ipilimumab .

Following the first 4 doses of the combination of nivolumab and ipilimumab, nivolumab monotherapy will again be given every 3 weeks at a dose of 360 mg for a maximum of 48 weeks. Patients may be dosed no less than 18 days from the previous dose of drug; and dosed up to 3 days after the scheduled date, if necessary.

ELIGIBILITY:
Inclusion Criteria-Part A:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

* Patients must have histologically confirmed advanced RCC (any histology). Collecting duct tumors and tumors originating from the renal pelvis or upper urinary tract are considered of urothelial origin and are excluded from this protocol.
* Patients must have at least one measurable site of disease, per RECIST 1.1, that has not been previously irradiated. If the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation.
* Archival tissue of a metastatic lesion obtained within 1 year prior to study registration (within 4 weeks preferred) and tumor tissue from nephrectomy is required if available. In addition to archival tissue of a metastatic lesion and nephrectomy, patients must have at least one site of disease (not including bone metastases) accessible for biopsy. If biopsy/resection of a new lesion or primary tumor and slow freezing of fresh tissue for single cell RNAseq study (as specified in the CLM) is not feasible, the subject is not eligible for the study. All biopsies must be core needle or excisional. Fine needle aspirate is not acceptable. NOTE: The tissue collected from a surgical resection or multiple core biopsies of either a metastatic lesion or primary tumor for the slow freezing of fresh tissue after the patient has signed consent for the study could also be used for collecting the FFPE specimens.
* ECOG performance status 0-2.
* Age ≥ 18 years.
* Have signed the current approved informed consent form.
* Patients must have adequate organ function within 14 days prior to study entry as evidenced by screening laboratory values that must meet the following criteria:

  * Hematological:

    * White blood cell (WBC) ≥ 2000/µL
    * Absolute Neutrophil Count (ANC) ≥ 1500/μL
    * Platelets (Plt) ≥ 100 x103/μL
    * Hemoglobin (Hgb) > 9.0 g/dL (with or without transfusion)
  * Renal:

    * Serum Creatinine ≤ 1.5 x ULN; if creatinine > 1.5, subject must demonstrate CrCl as outlined below.
    * Calculated creatinine clearance ≥ 40 mL/min using Cockcroft-Gault formula
  * Hepatic:

    * Bilirubin ≤ 1.5× upper limit of normal (ULN); Except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL
    * Aspartate aminotransferase (AST) ≤ 3 × ULN
    * Alanine aminotransferase (ALT) ≤ 3 × ULN
* Patients should not have received prior systemic therapy for metastatic RCC. Prior radiotherapy must have been completed at least 2 weeks prior to the administration of study drug. Patients must be 2 weeks from prior major surgery and 1 week from pre-treatment biopsy. Prior systemic adjuvant therapy (excluding with PD1 or CTLA4 pathway blockers) is allowed if treatment completed > 12 months previously.
* Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 5 months after the last dose of study drug. NOTE: Contraception is not required for male participants.
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) during screening for registration purposes. This pregnancy test should be repeated within 24 hours prior to the start of nivolumab. NOTE: "Women of childbearing potential" is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/ml.
* Women must not be breastfeeding.
* Be willing and able to comply with this protocol.

Exclusion Criteria:

* Patients are excluded if they have active brain metastases or leptomeningeal metastases. Subjects with brain metastases are eligible if metastases have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for 2 weeks of more after treatment is complete and within 28 days prior to the first dose of nivolumab administration. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.
* Patients with controlled brain metastases are allowed on protocol if they had solitary brain metastases that was surgically resected without recurrence or treated with SRS without progression x 4 weeks.
* Patients should be excluded if they have an active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* As there is potential for hepatic toxicity with nivolumab or nivolumab/ipilimumab combinations, drugs with a predisposition to hepatoxicity should be used with caution in patients treated with nivolumab-containing regimen
* Active infection requiring systemic therapy
* Has any other medical or personal condition that, in the opinion of the site investigator, may potentially compromise the safety or compliance of the patient, or may preclude the patient's successful completion of the clinical trial
* Patients should be excluded if they are positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
* Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Allergies and Adverse Drug Reaction

  * History of allergy to study drug components
  * History of severe hypersensitivity reaction to any monoclonal antibody
* Known additional malignancies within the past 3 years (excluding basal of squamous cell skin cancers, CIS or localized prostate cancer that has been treated or is being observed)

Inclusion/Exclusion Criteria- Part B

* Must meet eligibility criteria for initiation of Part A with the exception of being allowed to have prior nivolumab in Part A of this protocol
* Must have evidence of either RECIST 1.1 defined Disease Progression or Stable Disease 1 year after initiating nivolumab therapy
* Tumor biopsy prior to combination treatment is mandatory. If a biopsy/resection of a new lesion or primary tumor and slow freezing of fresh tissue for single cell RNAseq study (as specified in the CLM) is not feasible, the subject is not eligible for the study. All biopsies must be core needle or excisional. Fine needle aspirate is not acceptable.
* Must not have had a Grade ≥ 3 irAE on nivolumab monotherapy
* Must not have untreated brain metastases
* Must not have had major surgery or radiation therapy within 14 days of starting study treatment
* Must not have active autoimmune disease
* Must not have a concurrent medical condition requiring use of systemic corticosteroids with prednisone >10 mg per day
* Must not have had prior systemic therapy for Stage IV RCC (except for nivolumab as part of part A of this protocol)
* Prior solid organ or stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2025-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B. Atkins, MD, Study Chair — Hoosier Cancer Research Network
Locations (12):
- United States (12):
  - Yale University, Yale Cancer Center, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northwestern University Feinberg Schooll Of Medicine, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Beth Isreal Deaconess Medical Center, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Univeristy of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Atkins MB, Jegede OA, Haas NB, McDermott DF, Bilen MA, Stein M, Sosman JA, Alter R, Plimack ER, Ornstein MC, Hurwitz M, Peace DJ, Signoretti S, Denize T, Cimadamore A, Wu CJ, Braun D, Einstein D, Catalano PJ, Hammers H. Phase II study of nivolumab and salvage nivolumab/ipilimumab in treatment-naive patients with advanced non-clear cell renal cell carcinoma (HCRN GU16-260-Cohort B). J Immunother Cancer. 2023 Mar;11(3):e004780. doi: 10.1136/jitc-2022-004780. PMID 36948504
- [Derived] Atkins MB, Jegede OA, Haas NB, McDermott DF, Bilen MA, Stein M, Sosman JA, Alter R, Plimack ER, Ornstein M, Hurwitz M, Peace DJ, Signoretti S, Denize T, Cimadamore A, Wu CJ, Braun D, Einstein D, Catalano PJ, Hammers H. Phase II Study of Nivolumab and Salvage Nivolumab/Ipilimumab in Treatment-Naive Patients With Advanced Clear Cell Renal Cell Carcinoma (HCRN GU16-260-Cohort A). J Clin Oncol. 2022 Sep 1;40(25):2913-2923. doi: 10.1200/JCO.21.02938. Epub 2022 Apr 20. PMID 35442713
- See also: Hoosier Cancer Research Network Website — http://www.hoosiercancer.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Nivolumab and Salvage Nivolumab/Ipilimumab in Clear Cell RCC: All patients initiated treatment with nivolumab monotherapy (Part A). Those with progressive disease or stable disease at 48 weeks could receive a combination nivolumab/ipilimumab (Part B).
  PART A: Nivolumab
  Nivolumab 240 mg: Nivolumab 240 mg IV every 2 weeks x 6 then initial disease assessment.
  Nivolumab 360mg: Continue Nivolumab 360 mg IV every 3 weeks
  PART B: Nivolumab + Ipilimumab
  Ipilimumab 1mg/kg: Ipilimumab 1 mg/kg every 3 weeks x 4.
  Nivolumab 3mg/kg: In combination with Ipilimumab
  Nivolumab 360mg: Continue Nivolumab 360 mg IV every 3 weeks
- Cohort B: Nivolumab and Salvage Nivolumab/Ipilimumab in Non-clear Cell RCC: All patients initiated treatment with nivolumab monotherapy (Part A). Those with progressive disease or stable disease at 48 weeks could receive a combination nivolumab/ipilimumab (Part B).
  PART A: Nivolumab
  Nivolumab 240 mg: PART A Nivolumab 240 mg IV every 2 weeks x 6 then initial disease assessment
  Nivolumab 360mg: Continue Nivolumab 360 mg IV every 3 weeks
  PART B: Nivolumab + Ipilimumab
  Ipilimumab 1mg/kg: Ipilimumab 1 mg/kg every 3 weeks x 4
  Nivolumab 3mg/kg: In combination with Ipilimumab
  Nivolumab 360mg: Continue Nivolumab 360 mg IV every 3 weeks
Period: Overall Study
Arm/Group | Cohort A: Nivolumab and Salvage Nivolumab/Ipilimumab in Clear Cell RCC | Cohort B: Nivolumab and Salvage Nivolumab/Ipilimumab in Non-clear Cell RCC
Started | 128 | 36
Completed | 128 | 35
Not Completed | 0 | 1
Not completed — Not meeting inclusion criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Nivolumab and Salvage Nivolumab/Ipilimumab in Clear Cell RCC | Cohort B: Nivolumab and Salvage Nivolumab/Ipilimumab in Non-clear Cell RCC | Total
Number analyzed (Participants) | 128 | 35 | 163
Age, Continuous [Median (Full Range); unit: years] | 65 [32 to 86] | 63 [35 to 84] | 64 [32 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 4 | 40
  Male | 92 | 31 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 0 | 7
  Not Hispanic or Latino | 120 | 34 | 154
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 8 | 20
  White | 107 | 25 | 132
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 128 | 35 | 163
ECOG Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Dead:
  1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work, 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours.
  participants
    ECOG = 0 | 81 | 16 | 97
    ECOG = 1 | 46 | 17 | 63
    ECOG = 2 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: 1-year Progression Free Survival (PFS) Rate for ccRCC Patients
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  1-year Progression-Free Survival (PFS) Rate refers to the percentage of patients who have not experienced disease progression or death from any cause within one year of starting treatment. The 1-year PFS rate of nivolumab in treatment-naïve patients with clear cell renal cell carcinoma (ccRCC) was assessed according to tumor PD-L1 expression levels.
Time Frame: 1 year
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint progression-free survival for ccRCC patients was defined as all patients treated with nivolumab and has PD-L1 expression.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Cohort A Part A: Nivolumab Monotherapy in Clear Cell RCC: All patients initiated treatment with nivolumab monotherapy (Part A). Those with progressive disease or stable disease at 48 weeks could receive a combination nivolumab/ipilimumab (Part B).
  PART A: Nivolumab Nivolumab 240 mg: Nivolumab 240 mg IV every 2 weeks x 6 then initial disease assessment.
  Nivolumab 360mg: Continue Nivolumab 360 mg IV every 3 weeks
Arm/Group | Cohort A Part A: Nivolumab Monotherapy in Clear Cell RCC
Number analyzed (Participants) | 102
Percentage of participants
  PD-L1 0%: number analyzed (Participants) | 78
  PD-L1 0% | 34.6 [24.3 to 45.1]
  PD-L1 1-5%: number analyzed (Participants) | 13
  PD-L1 1-5% | 53.8 [24.8 to 76.0]
  PD-L1 5-20%: number analyzed (Participants) | 3
  PD-L1 5-20% | 33.3 [0.9 to 77.4]
  PD-L1 > 20%: number analyzed (Participants) | 8
  PD-L1 > 20% | 75 [31.5 to 93.1]

2. Secondary Outcome: Objective Response Rate for ccRCC Patients Treated With Nivolumab Monotherapy
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD. ORR = CR +PR Evaluate ORR for nivolumab in patients with treatment naïve clear cell renal cell carcinoma (ccRCC) based on PD-L1 expression.
Time Frame: Up to 39 Months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A Part A: Nivolumab Monotherapy in Clear Cell RCC
Number analyzed (Participants) | 102
Percentage of participants
  PD-L1 0%: number analyzed (Participants) | 78
  PD-L1 0% | 26.9 [17.5 to 38.2]
  PD-L1 1-5%: number analyzed (Participants) | 13
  PD-L1 1-5% | 53.8 [25.1 to 80.8]
  PD-L1 5-20%: number analyzed (Participants) | 3
  PD-L1 5-20% | 33.3 [0.8 to 90.6]
  PD-L1 > 20%: number analyzed (Participants) | 8
  PD-L1 > 20% | 75 [34.9 to 96.8]

3. Secondary Outcome: Objective Response Rate (ORR) for ccRCC Patients Treated With Nivolumab and Ipilimumab
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD. ORR = CR +PR. Evaluate ORR in combined nivolumab and ipilimumab therapy at the time of nivolumab failure for ccRCC patients based on PD-L1 expression.
Time Frame: Up to 39 Months
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint progression-free survival for Part B (treated with Nivolumab and Ipilimumab) ccRCC patients was defined as all patients who entered Part B and had PD-L1 expression.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Cohort A Part B: Nivolumab and Ipilimumab in Clear Cell RCC: All patients initiated treatment with nivolumab monotherapy (Part A). Those with progressive disease or stable disease at 48 weeks could receive a combination nivolumab/ipilimumab (Part B).
  PART B: Nivolumab + Ipilimumab Ipilimumab 1mg/kg: Ipilimumab 1 mg/kg every 3 weeks x 4. Nivolumab 3mg/kg: In combination with Ipilimumab Nivolumab 360mg: Continue Nivolumab 360 mg IV every 3 weeks
Arm/Group | Cohort A Part B: Nivolumab and Ipilimumab in Clear Cell RCC
Number analyzed (Participants) | 30
Percentage of participants
  PD-L1 0%: number analyzed (Participants) | 26
  PD-L1 0% | 7.7 [0.9 to 25.1]
  PD-L1 1-5%: number analyzed (Participants) | 3
  PD-L1 1-5% | 66.7 [9.4 to 99.2]
  PD-L1 5-20%: number analyzed (Participants) | 1
  PD-L1 5-20% | 0 [NA to NA] — Not enough events occur to calculate 95% confidence interval
  PD-L1 > 20%: number analyzed (Participants) | 0

4. Secondary Outcome: Clinical Activity for nccRCC Patients
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD. Clinical Activity = CR +PR+SD.
  Evaluate the clinical activity of nivolumab in patients with treatment naive nccRCC.
Time Frame: Up to 39 Months
Measure: Number; unit: Percentage of participants
Groups:
- Cohort B Part A: Nivolumab Monotherapy in Non Clear Cell RCC: All patients initiated treatment with nivolumab monotherapy (Part A). Those with progressive disease or stable disease at 48 weeks could receive a combination nivolumab/ipilimumab (Part B).
  PART A: Nivolumab Nivolumab 240 mg: PART A Nivolumab 240 mg IV every 2 weeks x 6 then initial disease assessment Nivolumab 360mg: Continue Nivolumab 360 mg IV every 3 weeks
Arm/Group | Cohort B Part A: Nivolumab Monotherapy in Non Clear Cell RCC
Number analyzed (Participants) | 35
Percentage of participants | 60

5. Secondary Outcome: 1-year Progression Free Survival (PFS) Rate for nccRCC Patients
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  1-year Progression-Free Survival (PFS) Rate refers to the percentage of patients who have not experienced disease progression or death from any cause within one year of starting treatment.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort B Part A: Nivolumab Monotherapy in Non Clear Cell RCC
Number analyzed (Participants) | 35
Percentage of participants | 25.4 [14.3 to 45]

6. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events will be assessed by the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) version 4.
Time Frame: Up to 28 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Nivolumab and Salvage Nivolumab/Ipilimumab in Clear Cell RCC | Cohort B: Nivolumab and Salvage Nivolumab/Ipilimumab in Non-clear Cell RCC
Number analyzed (Participants) | 128 | 35
Participants | 128 | 35

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored up to a maximum of 60 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored up to 28 months.
Groups:
- Cohort A Part B: Nivolumab/Ipilimumab in Clear Cell RCC: All patients initiated treatment with nivolumab monotherapy (Part A). Those with progressive disease or stable disease at 48 weeks could receive a combination nivolumab/ipilimumab (Part B).
  PART B: Nivolumab + Ipilimumab Ipilimumab 1mg/kg: Ipilimumab 1 mg/kg every 3 weeks x 4. Nivolumab 3mg/kg: In combination with Ipilimumab Nivolumab 360mg: Continue Nivolumab 360 mg IV every 3 weeks
- Cohort B Part A: Nivolumab Monotherapy in Non-clear Cell RCC: All patients initiated treatment with nivolumab monotherapy (Part A). Those with progressive disease or stable disease at 48 weeks could receive a combination nivolumab/ipilimumab (Part B).
  PART A: Nivolumab Nivolumab 240 mg: PART A Nivolumab 240 mg IV every 2 weeks x 6 then initial disease assessment Nivolumab 360mg: Continue Nivolumab 360 mg IV every 3 weeks
- Cohort B Part B: Nivolumab/Ipilimumab in Non-clear Cell RCC: All patients initiated treatment with nivolumab monotherapy (Part A). Those with progressive disease or stable disease at 48 weeks could receive a combination nivolumab/ipilimumab (Part B).
  PART B: Nivolumab + Ipilimumab Ipilimumab 1mg/kg: Ipilimumab 1 mg/kg every 3 weeks x 4 Nivolumab 3mg/kg: In combination with Ipilimumab Nivolumab 360mg: Continue Nivolumab 360 mg IV every 3 weeks
Arm/Group | Cohort A Part A: Nivolumab Monotherapy in Clear Cell RCC | Cohort A Part B: Nivolumab/Ipilimumab in Clear Cell RCC | Cohort B Part A: Nivolumab Monotherapy in Non-clear Cell RCC | Cohort B Part B: Nivolumab/Ipilimumab in Non-clear Cell RCC
All-Cause Mortality (participants affected / at risk) | 38/128 | 28/40 | 11/35 | 15/17
Serious Adverse Events (participants affected / at risk) | 41/128 | 19/40 | 8/35 | 5/17
Other Adverse Events (participants affected / at risk) | 127/128 | 38/40 | 34/35 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A Part A: Nivolumab Monotherapy in Clear Cell RCC (N=128) | Cohort A Part B: Nivolumab/Ipilimumab in Clear Cell RCC (N=40) | Cohort B Part A: Nivolumab Monotherapy in Non-clear Cell RCC (N=35) | Cohort B Part B: Nivolumab/Ipilimumab in Non-clear Cell RCC (N=17)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALLERGIC REACTION (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ANEMIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
CARDIAC DISORDERS - OTHER, SPECIFY (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COGNITIVE DISTURBANCE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
CONFUSION (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CREATININE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEATH NOS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DELUSIONS (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
EDEMA CEREBRAL (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ENCEPHALITIS INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FACIAL NERVE DISORDER (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FEVER (General disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
HEART FAILURE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
LUNG INFECTION (Infections and infestations) | 4 (5) | 0 (0) | 0 (0) | 1 (1)
MENINGISMUS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
MYOCARDITIS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 1 (2) | 0 (0)
RETROPERITONEAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEIZURE (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 2 (2) | 1 (1) | 1 (2) | 0 (0)
SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
STEVENS-JOHNSON SYNDROME (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
STROKE (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
TRANSIENT ISCHEMIC ATTACKS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIAC TROPONIN I INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GALLBLADDER OBSTRUCTION (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEPATOBILIARY DISORDERS - OTHER, SPECIFY (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LIPASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MYOSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SERUM AMYLASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BRONCHOPULMONARY HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EDEMA LIMBS (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
ESOPHAGEAL HEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TUMOR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASCITES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUDDEN DEATH NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A Part A: Nivolumab Monotherapy in Clear Cell RCC (N=128) | Cohort A Part B: Nivolumab/Ipilimumab in Clear Cell RCC (N=40) | Cohort B Part A: Nivolumab Monotherapy in Non-clear Cell RCC (N=35) | Cohort B Part B: Nivolumab/Ipilimumab in Non-clear Cell RCC (N=17)
ABDOMINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 19 (23) | 5 (5) | 6 (8) | 4 (7)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 3 (3) | 3 (4) | 0 (0) | 0 (0)
AGITATION (Psychiatric disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 23 (37) | 5 (7) | 5 (7) | 2 (4)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 31 (49) | 5 (6) | 8 (11) | 4 (6)
ALLERGIC REACTION (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 2 (2) | 1 (1) | 0 (0)
AMNESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANEMIA (Blood and lymphatic system disorders) | 34 (68) | 9 (14) | 14 (26) | 6 (12)
ANOREXIA (Metabolism and nutrition disorders) | 14 (17) | 9 (14) | 4 (4) | 2 (3)
ANXIETY (Psychiatric disorders) | 10 (12) | 1 (1) | 3 (3) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 31 (45) | 1 (1) | 1 (1) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 7 (9) | 0 (0) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 21 (31) | 4 (6) | 5 (6) | 3 (4)
ATAXIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 30 (42) | 4 (4) | 8 (9) | 7 (7)
BLOATING (Gastrointestinal disorders) | 5 (5) | 1 (2) | 0 (0) | 1 (1)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (Blood and lymphatic system disorders) | 14 (22) | 0 (0) | 3 (3) | 2 (2)
BLOOD BILIRUBIN INCREASED (Investigations) | 9 (14) | 3 (3) | 1 (6) | 0 (0)
BLURRED VISION (Eye disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 4 (8) | 1 (1) | 0 (0) | 1 (1)
BREAST PAIN (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
BRONCHIAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRUISING (Injury, poisoning and procedural complications) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CARDIAC DISORDERS - OTHER, SPECIFY (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
CARDIAC TROPONIN I INCREASED (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
CARDIAC TROPONIN T INCREASED (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
CHEST PAIN - CARDIAC (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
CHILLS (General disorders) | 7 (11) | 3 (3) | 1 (2) | 0 (0)
CHOLESTEROL HIGH (Investigations) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (4)
COLITIS (Gastrointestinal disorders) | 5 (9) | 1 (1) | 0 (0) | 1 (2)
CONFUSION (Psychiatric disorders) | 3 (6) | 0 (0) | 0 (0) | 1 (1)
CONGENITAL, FAMILIAL AND GENETIC DISORDERS - OTHER, SPECIFY (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 26 (30) | 5 (6) | 7 (10) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 47 (66) | 10 (16) | 7 (8) | 3 (3)
CPK INCREASED (Investigations) | 11 (19) | 1 (5) | 2 (3) | 2 (2)
CREATININE INCREASED (Investigations) | 44 (82) | 14 (20) | 11 (16) | 3 (3)
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 5 (8) | 2 (2) | 0 (0) | 0 (0)
DELIRIUM (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 5 (5) | 1 (1) | 1 (1) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 41 (80) | 11 (23) | 6 (8) | 4 (6)
DIZZINESS (Nervous system disorders) | 17 (20) | 5 (9) | 5 (7) | 1 (2)
DRY EYE (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 8 (10) | 6 (6) | 2 (2) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 12 (15) | 1 (1) | 3 (4) | 0 (0)
DUODENAL HEMORRHAGE (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 4 (4) | 2 (3) | 0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 6 (7) | 0 (0) | 2 (2) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 22 (26) | 8 (9) | 6 (7) | 2 (3)
EAR AND LABYRINTH DISORDERS - OTHER, SPECIFY (Ear and labyrinth disorders) | 4 (5) | 0 (0) | 1 (1) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
EDEMA LIMBS (General disorders) | 11 (15) | 4 (4) | 5 (6) | 0 (0)
ENCEPHALITIS INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ENDOCRINE DISORDERS - OTHER, SPECIFY (Endocrine disorders) | 4 (6) | 2 (3) | 0 (0) | 1 (1)
ENTEROCOLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
EXTERNAL EAR INFLAMMATION (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EXTRAPYRAMIDAL DISORDER (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EYE DISORDERS - OTHER, SPECIFY (Eye disorders) | 8 (10) | 1 (2) | 0 (0) | 0 (0)
FACIAL NERVE DISORDER (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FACIAL PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 4 (11) | 1 (1) | 2 (2) | 0 (0)
FATIGUE (General disorders) | 63 (88) | 17 (26) | 16 (25) | 8 (10)
FEVER (General disorders) | 6 (6) | 3 (4) | 3 (5) | 2 (4)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 1 (2) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FLOATERS (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FLU LIKE SYMPTOMS (General disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
FLUSHING (Vascular disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 5 (6) | 3 (3) | 2 (2) | 3 (3)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 10 (13) | 2 (5) | 2 (2) | 2 (2)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 16 (21) | 1 (1) | 2 (3) | 1 (1)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (1) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 29 (41) | 4 (4) | 4 (5) | 3 (4)
HEARING IMPAIRED (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
HEART FAILURE (Cardiac disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
HEMATOMA (Vascular disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
HEMATURIA (Renal and urinary disorders) | 8 (11) | 2 (6) | 2 (2) | 1 (1)
HEMOGLOBIN INCREASED (Investigations) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
HEMORRHOIDAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEMORRHOIDS (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
HEPATOBILIARY DISORDERS - OTHER, SPECIFY (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
HOT FLASHES (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 10 (12) | 5 (9) | 0 (0) | 0 (0)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 24 (54) | 3 (5) | 3 (7) | 2 (3)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
HYPERKALEMIA (Metabolism and nutrition disorders) | 18 (43) | 5 (6) | 5 (10) | 3 (4)
HYPERNATREMIA (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 36 (117) | 11 (28) | 5 (14) | 2 (9)
HYPERTHYROIDISM (Endocrine disorders) | 4 (5) | 2 (3) | 1 (1) | 1 (1)
HYPERURICEMIA (Metabolism and nutrition disorders) | 29 (43) | 3 (4) | 7 (15) | 6 (10)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 14 (20) | 6 (8) | 6 (8) | 0 (0)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 8 (12) | 2 (2) | 1 (1) | 0 (0)
HYPOKALEMIA (Metabolism and nutrition disorders) | 5 (7) | 5 (10) | 2 (5) | 2 (2)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1) | 3 (5) | 0 (0) | 0 (0)
HYPONATREMIA (Metabolism and nutrition disorders) | 22 (37) | 3 (3) | 2 (5) | 1 (1)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 8 (18) | 1 (1) | 2 (2) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 24 (29) | 5 (7) | 1 (1) | 4 (6)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 7 (15) | 2 (2) | 1 (1) | 2 (2)
INFUSION RELATED REACTION (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
INR INCREASED (Investigations) | 1 (4) | 1 (1) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 20 (23) | 0 (0) | 0 (0) | 0 (0)
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
IRRITABILITY (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LETHARGY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LIP INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
LIPASE INCREASED (Investigations) | 33 (98) | 12 (34) | 2 (3) | 2 (11)
LOCALIZED EDEMA (General disorders) | 7 (7) | 1 (1) | 2 (2) | 0 (0)
LUNG INFECTION (Infections and infestations) | 6 (7) | 0 (0) | 1 (1) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 3 (6) | 2 (2) | 1 (1) | 0 (0)
MALAISE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MANIA (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MEMORY IMPAIRMENT (Nervous system disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
MENINGISMUS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
MITRAL VALVE DISEASE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUCOSAL INFECTION (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 7 (8) | 1 (1) | 2 (3) | 2 (2)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
MUSCLE WEAKNESS UPPER LIMB (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 23 (30) | 6 (6) | 4 (6) | 4 (6)
MYALGIA (Musculoskeletal and connective tissue disorders) | 13 (19) | 1 (1) | 2 (2) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYOSITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
NAIL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 23 (31) | 5 (5) | 3 (3) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 32 (40) | 10 (16) | 8 (11) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 6 (9) | 1 (1) | 0 (0) | 1 (1)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 1 (1) | 1 (1) | 0 (0)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 5 (5) | 2 (2) | 1 (3) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 3 (7) | 0 (0) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 4 (5) | 2 (2) | 1 (1) | 2 (4)
OBESITY (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ORAL DYSESTHESIA (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ORAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTITIS EXTERNA (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
PAIN (General disorders) | 16 (19) | 7 (8) | 4 (4) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 27 (44) | 7 (10) | 4 (5) | 3 (6)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PALMAR-PLANTAR ERYTHRODYSESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
PALPITATIONS (Cardiac disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
PAPULOPUSTULAR RASH (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
PARESTHESIA (Nervous system disorders) | 4 (6) | 1 (2) | 2 (2) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
PERICARDITIS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 12 (12) | 1 (1) | 1 (1) | 0 (0)
PHLEBITIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 9 (22) | 0 (0) | 1 (2) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 1 (1) | 0 (0) | 0 (0)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (2) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 1 (3) | 0 (0)
PROSTATIC OBSTRUCTION (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 45 (61) | 11 (18) | 6 (6) | 4 (5)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 43 (72) | 13 (25) | 10 (13) | 10 (15)
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
REPRODUCTIVE SYSTEM AND BREAST DISORDERS - OTHER, SPECIFY (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 1 (1) | 1 (1) | 0 (0)
RHINITIS INFECTIVE (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
SERUM AMYLASE INCREASED (Investigations) | 27 (68) | 8 (19) | 5 (6) | 1 (3)
SINUS BRADYCARDIA (Cardiac disorders) | 4 (5) | 0 (0) | 1 (1) | 1 (1)
SINUS PAIN (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 3 (6) | 2 (2) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 25 (50) | 4 (8) | 7 (12) | 0 (0)
SKIN ATROPHY (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN INFECTION (Infections and infestations) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0) | 1 (1) | 0 (0)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 0 (0) | 0 (0) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
STROKE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SURGICAL AND MEDICAL PROCEDURES - OTHER, SPECIFY (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
THROMBOEMBOLIC EVENT (Vascular disorders) | 3 (4) | 4 (6) | 1 (2) | 2 (2)
TINNITUS (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
TOXIC EPIDERMAL NECROLYSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
TUMOR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 15 (19) | 1 (1) | 3 (5) | 0 (0)
URINARY FREQUENCY (Renal and urinary disorders) | 7 (9) | 0 (0) | 0 (0) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 9 (13) | 1 (2) | 1 (1) | 1 (1)
URINARY TRACT PAIN (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
URINARY URGENCY (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
URINE DISCOLORATION (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UVEITIS (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
VAGINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VASCULAR DISORDERS - OTHER, SPECIFY (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
VASOVAGAL REACTION (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 9 (13) | 8 (10) | 4 (5) | 0 (0)
WATERING EYES (Eye disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
WEIGHT GAIN (Investigations) | 11 (17) | 4 (5) | 1 (1) | 0 (0)
WEIGHT LOSS (Investigations) | 16 (25) | 11 (17) | 5 (5) | 5 (8)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
WHITE BLOOD CELL DECREASED (Investigations) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
BULLOUS DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
ELECTROCARDIOGRAM QT CORRECTED INTERVAL PROLONGED (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
EYE PAIN (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EYELID FUNCTION DISORDER (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FECAL INCONTINENCE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 1 (1) | 2 (2)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
STOMACH PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALKALOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AUTOIMMUNE DISORDER (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
BRONCHOPULMONARY HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
CONJUNCTIVITIS (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GENITAL EDEMA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GLAUCOMA (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GYNECOMASTIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAPTOGLOBIN DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERPARATHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOICE ALTERATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INJECTION SITE REACTION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/09/NCT03117309/Prot_SAP_000.pdf